CLINICAL TRIAL: NCT01350076
Title: Liberal VS Goal-directed Intraoperative Fluid Therapy in Pediatric Patients
Brief Title: Liberal Versus Goal-directed Intraoperative Fluid Therapy in Pediatric Patients
Acronym: GDT
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mahidol University (Other)
Responsible Party: Suwannee Suraseranivongse, Faculty of Medicine Siriraj Hospital, Mahidol University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Si 511/2010
Record Dates: First submitted 2011-03-30; First posted 2011-05-09 (Estimated); Last update posted 2011-05-09 (Estimated); Status verified 2011-05

CONDITIONS: Adverse Anesthesia Outcome
Keywords: intraoperative fluid; pediatric; goal directed therapy; pediatric with major abdominal surgery; ASA less than or equal to 3; Duration of surgery less than 2 hours; Body weight more than or equal to 15 kg
MeSH Terms: interventions — Crystalloid Solutions

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- control group (Active Comparator): Control group will receive conventional liberal fluid regimen with crystalloid Liberal fluid regimen = Maintenance fluid + fasting fluid + dehydration + third space loss Maintenance fluid = (4X BW 1-10 kg) + (2X1BW11-20 kg) + (1X BW 0ver 21 kg) Fasting fluid = maintenance fluid X fasting duration
  Interventions: Drug: conventional liberal fluid regimen
- study group (Experimental): Study group will receive restricted fluid regimen (the same as control group except third space replacement) plus goal directed fluid therapy to maintain adequate CO guided by USCOM as shown in diagram (figure 1).
  Figure 1 goal directed fluid therapy SVV = Stroke volume variation SVI = Stroke volume index CI = Cardiac index
  Interventions: Drug: restricted fluid regimen

INTERVENTIONS:
Drug: conventional liberal fluid regimen — Control group will receive conventional liberal fluid regimen with crystalloid Liberal fluid regimen = Maintenance fluid + fasting fluid + dehydration + third space loss Maintenance fluid = (4X BW 1-10 kg) + (2X1BW11-20 kg) + (1X BW 0ver 21 kg) Fasting fluid = maintenance fluid X fasting duration
  Other Names: crystalloid
  Arms: control group
Drug: restricted fluid regimen — Study group will receive restricted fluid regimen (the same as control group except third space replacement) plus goal directed fluid therapy to maintain adequate CO guided by USCOM as shown in diagram (figure 1).
  Figure 1 goal directed fluid therapy SVV = Stroke volume variation SVI = Stroke volume index CI = Cardiac index
  Other Names: crystalloid
  Arms: study group

SUMMARY:
The objectives of this study are 1) to investigate the influence of different fluid regimen (Liberal regimen versus Goal directed therapy regimen) on postoperative outcome such as weight gain, delayed gut function recovery, pneumonia and 2) to ascertain the reliability of USCOM monitoring using serum lactate and base deficit as control parameters.

DETAILED DESCRIPTION:
Liberal regimen = maintenance fluid(4/2/1) + deficit fluid + replacement of third space loss (>,=10ml/kg/h) Goal directed therapy regimen = maintenance fluid + deficit fluid + fluid replaced by hemodynamic monitoring guided.

ELIGIBILITY:
Inclusion Criteria:

* Body weight < 15 kg
* Under going major abdominal surgery such as tumor removal, gut obstruction, pull through, etc. under general anesthesia and invasive arterial pressure monitoring if justified
* ASA < or = 3
* Duration of surgery > or = 2 hours

Exclusion Criteria:

* Cardiopulmonary disease
* Renal insufficiency
* Intraoperative complications such as massive bleeding, severe hypotension, prolonged need for mandatory ventilation
* reoperation

Ages: 1 Minute to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2011-10; Primary Completion 2013-06 (Estimated); Study Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with 5% postoperative weight gain between control group and study group | 24 hours
  Body weight

SECONDARY OUTCOMES:
Postoperative morbidity | 4 days
  Postoperative morbidity: lung (new postoperative infiltration), prolonged ileus means inability to feed in postoperative day 4, kidney ( increase BUN, Cr), tissue hypoxia (wound infection, anastomotic leakage)
Amount of intraoperative fluid | 1 day
  Amount of intraoperative fluid

CONTACTS AND LOCATIONS:
Overall Officials: Suwannee Suraseranivongse, MD, Principal Investigator — Mahidol University
Locations (1):
- Siriraj Hospital, Bangkok, Bangkok, Thailand